CLINICAL TRIAL: NCT01041638
Title: A Comprehensive Safety Trial of Chimeric Antibody 14.18 (Ch14.18) With GM-CSF, IL-2 and Isotretinoin in High-Risk Neuroblastoma Patients Following Myeloablative Therapy
Brief Title: Monoclonal Antibody Ch14.18, Sargramostim, Aldesleukin, and Isotretinoin After Autologous Stem Cell Transplant in Treating Patients With Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01997; NCI-2011-01997 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ANBL0931; ANBL0931; CDR0000662673; ANBL0931 (Other: Children's Oncology Group); ANBL0931 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2009-12-31; First posted 2010-01-01 (Estimated); Results first posted 2015-02-19 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-06

CONDITIONS: High Risk Neuroblastoma
MeSH Terms: interventions — aldesleukin; dinutuximab; Isotretinoin; sargramostim; Colony-Stimulating Factors

ARMS (1):
- Treatment (Ch14.18, GM-CSF, IL-2, isotretinoin) (Experimental): Patients receive sargramostim SC or IV over 2 hours on days 0-13 of courses 1, 3, and 5; monoclonal antibody Ch14.18 IV over 10 hours on days 3-6 of courses 1, 3, and 5 and on days 7-10 of courses 2 and 4; and isotretinoin PO BID on days 11-24 of course 1, on days 14-27 of courses 2, 4, and 6, and on days 10-23 of courses 3 and 5. Patients also receive aldesleukin IV continuously on days 0-3 and on days 7-10 of courses 2 and 4. Treatment repeats every 24-32 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Aldesleukin; Other: Diagnostic Laboratory Biomarker Analysis; Biological: Dinutuximab; Drug: Isotretinoin; Biological: Sargramostim

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Biological: Dinutuximab — Given IV
  Other Names: Ch 14.18UTC; Ch14.18; MOAB Ch14.18; monoclonal antibody Ch14.18; Unituxin
Drug: Isotretinoin — Given PO
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Absorica; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Myorisan; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret; ZENATANE
Biological: Sargramostim — Given IV or SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
This phase III trial is studying the side effects of giving monoclonal antibody Ch14.18 together with sargramostim, aldesleukin, and isotretinoin after autologous stem cell transplant in treating patients with neuroblastoma. Monoclonal antibodies, such as Ch14.18, may find tumor cells and help kill them. Colony-stimulating factors, such as sargramostim, may increase the number of immune cells found in bone marrow or peripheral blood. Aldesleukin may stimulate the white blood cells to kill tumor cells. Isotretinoin may help neuroblastoma cells become more like normal cells, and to grow and spread more slowly. Giving monoclonal antibody Ch14.18 with sargramostim, aldesleukin, and isotretinoin after autologous stem cell transplant may be an effective treatment for neuroblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To comprehensively define the safety profile of ch14.18 when administered with cytokines and isotretinoin in high-risk neuroblastoma patients after autologous stem cell transplant (ASCT).

SECONDARY OBJECTIVES:

I. To further describe and refine the event-free survival (EFS) and overall survival (OS) estimates and baseline characteristics for subjects receiving chl4.18 + cytokines + isotretinoin.

II. To further describe the safety and toxicity of chl4.18 + cytokines + isotretinoin with focus on: a) number of courses delivered per patient; b) number of dose reductions or stoppage (ch14.18 and/or interleukin [IL]-2 [aldesleukin]); and c) number of toxic deaths.

III. To further describe the immune reconstitution of patients following ASCT, based on laboratory data obtained just prior to, during, and after treatment with this regimen.

IV. To obtain correlative laboratory data to evaluate and describe mechanisms related to response, toxicity of immune activation, and allergic phenomena.

OUTLINE:

Patients receive sargramostim subcutaneously (SC) or intravenously (IV) over 2 hours on days 0-13 of courses 1, 3, and 5; monoclonal antibody Ch14.18 IV over 10 hours on days 3-6 of courses 1, 3, and 5 and on days 7-10 of courses 2 and 4; and isotretinoin orally (PO) twice daily (BID) on days 11-24 of course 1, on days 14-27 of courses 2, 4, and 6, and on days 10-23 of courses 3 and 5. Patients also receive aldesleukin IV continuously on days 0-3 and on days 7-10 of courses 2 and 4. Treatment repeats every 24-32 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 1 year, every 6 months for 4 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be diagnosed with neuroblastoma, and categorized as high-risk at the time of diagnosis
* At pre-ASCT evaluation, patients must meet the International Neuroblastoma Response Criteria (INRC) for complete response (CR), very good partial response (VGPR), or partial response (PR) for primary site, soft tissue metastases and bone metastases; patients who meet those criteria must also meet the protocol specified criteria for bone marrow response as outlined below: =< 10% tumor (of total nucleated cellular content) seen on any specimen from a bilateral bone marrow aspirate/biopsy; patients who have no tumor seen on the prior bone marrow, and then have =< 10% tumor on any of the bilateral marrow aspirate/biopsy specimens done at pre-ASCT and/or pre-enrollment evaluation will also be eligible; (Note that, per INRC, this would have been defined as an "overall" response of progressive disease [PD])
* Prior to enrollment on ANBL0931, a determination of residual disease must be performed (tumor imaging studies including metaiodobenzylguanidine [MIBG] scan, computed tomography [CT] or magnetic resonance imaging [MRI], bone marrow aspiration and biopsy); this disease assessment is required for eligibility, and should be done preferably within 2 weeks but must be done within a maximum of 4 weeks before enrollment

  * Patients with residual disease are eligible; biopsy is not required
  * Patients must not have progressive disease except for protocol specified bone marrow response
* All patients must have completed therapy including intensive induction chemotherapy followed by ASCT and radiotherapy to be eligible; radiotherapy may be waived for patients who either had a small adrenal mass which was completely resected upfront, or who never had an identifiable primary tumor
* No more than 9 months from the date of starting the first induction chemotherapy after diagnosis to the date of ASCT except for the rare occasions as noted below; for tandem ASCT patients, this will be the date of the FIRST stem cell infusion; Exception: for those who are initially diagnosed as non-high risk neuroblastoma, but later converted (and/ or relapsed) to high risk neuroblastoma, the 9 months restriction should start from the date of induction therapy for high risk neuroblastoma (not from the initial induction therapy for non-high risk disease), to the date of ASCT
* Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age; required patients must have a Lansky or Karnofsky performance scale score of >= 50%
* Patients must have a life expectancy of >= 2 months (8 weeks)
* Total absolute phagocyte count (APC = neutrophils + monocytes) is at least 1000/uL
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 month to < 6 months: 0.4 mg/dL
  * 6 months to < 1 year: 0.5 mg/dL
  * 1 to < 2 years: 0.6 mg/dL
  * 2 to < 6 years: 0.8 mg/dL
  * 6 to < 10 years: 1 mg/dL
  * 10 to < 13 years: 1.2 mg/dL
  * 13 to < 16 years: 1.5 mg/dL (male), 1.4 mg/dL (female)
  * >= 16 years: 1.7 mg/dL (male), 1.4 mg/dL (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 5 x upper limit of normal (ULN) for age
* SOS (sinusoidal obstruction syndrome, formerly known as veno-occlusive disease [VOD]), if present, should be stable or improving
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 55% by radionuclide angiography
* No evidence of dyspnea at rest
* If pulmonary function tests (PFTs) are performed, forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) > 60% by pulmonary function test
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* Central nervous system (CNS) toxicity < grade 2

Exclusion Criteria:

* Females of childbearing potential must have a negative pregnancy test
* Patients of childbearing potential must agree to use an effective birth control method
* Female patients who are lactating must agree to stop breast-feeding
* Patients must not have received prior anti-GD2 antibody therapy
* Patients must not have received prior vaccine therapy administered as treatment of neuroblastoma not routine infectious disease vaccinations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-12-21 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet F Ozkaynak, Principal Investigator — Children's Oncology Group
Locations (32):
- United States (32):
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Chimeric Antibody 14.18 With GM-CSF, IL-2 and Isotretinoin: Patients receive sargramostim subcutaneously or IV over 2 hours on days 0-13 of courses 1, 3, and 5 (dose: 250 micrograms/m²/dose); monoclonal antibody Ch14.18 IV over 10 hours on days 3-6 of courses 1, 3, and 5 and on days 7-10 of courses 2 and 4 (dose: 25 mg/m2/dose); and oral isotretinoin twice daily on days 11-24 of course 1, on days 14-27 of courses 2, 4, and 6, and on days 10-23 of courses 3 and 5 (Weight based dosage: > 12 kg: 80 mg/m2/dose BID; total daily dose 160 mg/m2/day, divided BID. ≤ 12 kg: 2.67 mg/kg/dose BID; total daily dose is 5.33 mg/kg/day, divided BID. Round dose up to the nearest 10 mg). Patients also receive aldesleukin IV continuously on days 0-3 and on days 7-10 of courses 2 and 4 (actual dosage is body surface area based and varies by course). Treatment repeats every 24-32 days for 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Chimeric Antibody 14.18 With GM-CSF, IL-2 and Isotretinoin
Started | 105
Completed | 78
Not Completed | 27
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Lack of Efficacy | 7
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 11

BASELINE CHARACTERISTICS:
Arm/Group | Chimeric Antibody 14.18 With GM-CSF, IL-2 and Isotretinoin
Number analyzed (Participants) | 105
Age, Continuous [Median (Full Range); unit: years] | 4.1 [1.1 to 27.5]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 103
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 82
  More than one race | 0
  Unknown or Not Reported | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 87
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 105

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Experienced a Significant (CTC Grade 3-5) Nonhematologic Toxicity of Interest (Pain, Hypotension, Allergic Reactions, Capillary Leak Syndrome, or Fever).
Description: Designed to collect comprehensive safety/toxicity data, as well as additional efficacy data for the immunotherapy. To address the primary objective, descriptive analyses summarizing the number and type of AEs will be performed. The percentage of patients reporting each unacceptable (Grade 3 or higher) CTC toxicity code, tabulated by course, are reported.
Time Frame: Up to 6 courses of therapy
Population: There was one patient that did not receive treatment, represented on the baseline form as "withdrawal by patient", not included in outcome measure tabulation.
Measure: Number; unit: percentage of participants
Arm/Group | Chimeric Antibody 14.18 With GM-CSF, IL-2 and Isotretinoin
Number analyzed (Participants) | 104
percentage of participants
  Abdominal pain (10300), course 1 | 17.3077
  Abdominal pain (10300), course 2 | 5.0000
  Abdominal pain (10300), course 3 | 6.1224
  Abdominal pain (10300), course 4 | 4.4444
  Abdominal pain (10300), course 5 | 5.6818
  Abdominal pain (10300), course 6 | 0.00000
  Allergic reaction (12000), Course 1 | 1.92308
  Allergic reaction (12000), Course 2 | 5.00000
  Allergic reaction (12000), Course 3 | 3.06122
  Allergic reaction (12000), Course 4 | 2.22222
  Allergic reaction (12000), Course 5 | 1.13636
  Allergic reaction (12000), Course 6 | 0.00000
  Anal pain (12800), Course 1 | 0.00000
  Anal pain (12800), Course 2 | 1.00000
  Anal pain (12800), Course 3 | 0.00000
  Anal pain (12800), Course 4 | 0.00000
  Anal pain (12800), Course 5 | 0.00000
  Anal pain (12800), Course 6 | 0.00000
  Anaphylaxis (13100), Course 1 | 0.96154
  Anaphylaxis (13100), Course 2 | 4.00000
  Anaphylaxis (13100), Course 3 | 1.02041
  Anaphylaxis (13100), Course 4 | 3.33333
  Anaphylaxis (13100), Course 5 | 1.13636
  Anaphylaxis (13100), Course 6 | 0.00000
  Back pain (16200), Course 1 | 4.80769
  Back pain (16200), Course 2 | 5.00000
  Back pain (16200), Course 3 | 3.06122
  Back pain (16200), Course 4 | 3.33333
  Back pain (16200), Course 5 | 4.54545
  Back pain (16200), Course 6 | 0.00000
  Capillary leak syndrome (19800) - Course 1 | 0.96154
  Capillary leak syndrome (19800) - Course 2 | 4.00000
  Capillary leak syndrome (19800) - Course 3 | 0.00000
  Capillary leak syndrome (19800) - Course 4 | 2.22222
  Capillary leak syndrome (19800) - Course 5 | 0.00000
  Capillary leak syndrome (19800) - Course 6 | 0.00000
  Chest wall pain (21400) - Course 1 | 0.00000
  Chest wall pain (21400) - Course 2 | 0.00000
  Chest wall pain (21400) - Course 3 | 1.02041
  Chest wall pain (21400) - Course 4 | 0.00000
  Chest wall pain (21400) - Course 5 | 1.13636
  Chest wall pain (21400) - Course 6 | 0.00000
  Fever (33900) - Course 1 | 21.1538
  Fever (33900) - Course 2 | 58.0000
  Fever (33900) - Course 3 | 6.1224
  Fever (33900) - Course 4 | 31.1111
  Fever (33900) - Course 5 | 4.5455
  Fever (33900) - Course 6 | 1.2346
  Flank pain (34200) - Course 1 | 0.96154
  Flank pain (34200) - Course 2 | 0.00000
  Flank pain (34200) - Course 3 | 0.00000
  Flank pain (34200) - Course 4 | 0.00000
  Flank pain (34200) - Course 5 | 0.00000
  Flank pain (34200) - Course 6 | 0.00000
  Hypotension (43600) - Course 1 | 9.6154
  Hypotension (43600) - Course 2 | 17.0000
  Hypotension (43600) - Course 3 | 4.0816
  Hypotension (43600) - Course 4 | 14.4444
  Hypotension (43600) - Course 5 | 7.9545
  Hypotension (43600) - Course 6 | 0.00000
  Neck pain (57800) - Course 1 | 0.96154
  Neck pain (57800) - Course 2 | 3.00000
  Neck pain (57800) - Course 3 | 0.00000
  Neck pain (57800) - Course 4 | 0.00000
  Neck pain (57800) - Course 5 | 1.13636
  Neck pain (57800) - Course 6 | 0.00000
  Non-cardiac chest pain (58600) - Course 1 | 0.96154
  Non-cardiac chest pain (58600) - Course 2 | 0.00000
  Non-cardiac chest pain (58600) - Course 3 | 0.00000
  Non-cardiac chest pain (58600) - Course 4 | 0.00000
  Non-cardiac chest pain (58600) - Course 5 | 0.00000
  Non-cardiac chest pain (58600) - Course 6 | 0.00000
  Pain (60600) - Course 1 | 23.0769
  Pain (60600) - Course 2 | 16.0000
  Pain (60600) - Course 3 | 13.2653
  Pain (60600) - Course 4 | 20.0000
  Pain (60600) - Course 5 | 11.3636
  Pain (60600) - Course 6 | 1.2346
  Pain in extremity (60700) - Course 1 | 4.80769
  Pain in extremity (60700) - Course 2 | 4.00000
  Pain in extremity (60700) - Course 3 | 3.06122
  Pain in extremity (60700) - Course 4 | 6.66667
  Pain in extremity (60700) - Course 5 | 2.27273
  Pain in extremity (60700) - Course 6 | 1.23457
  Peripheral sensory neuropathy (64100) - Course 1 | 0.96154
  Peripheral sensory neuropathy (64100) - Course 2 | 0.00000
  Peripheral sensory neuropathy (64100) - Course 3 | 1.02041
  Peripheral sensory neuropathy (64100) - Course 4 | 0.00000
  Peripheral sensory neuropathy (64100) - Course 5 | 0.00000
  Peripheral sensory neuropathy (64100) - Course 6 | 0.00000

2. Secondary Outcome: Event-free Survival (EFS)
Description: Event-free Survival (EFS) for all eligible patients enrolled on the study
Time Frame: From enrollment until the first occurrence of relapse, progressive disease, secondary malignancy, or death, or until last contact if no event occurred, up to 3 years
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Chimeric Antibody 14.18 With GM-CSF, IL-2 and Isotretinoin
Number analyzed (Participants) | 105
percentage | 67.6 [58.2 to 77.0]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) for all eligible patients enrolled on the study
Time Frame: From enrollment until death, or until last contact with the patient, up to 3 years
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Chimeric Antibody 14.18 With GM-CSF, IL-2 and Isotretinoin
Number analyzed (Participants) | 105
percentage | 79.1 [70.9 to 87.3]

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs.
Arm/Group | Chimeric Antibody 14.18 With GM-CSF, IL-2 and Isotretinoin
Serious Adverse Events (participants affected / at risk) | 103/104
Other Adverse Events (participants affected / at risk) | 104/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chimeric Antibody 14.18 With GM-CSF, IL-2 and Isotretinoin (N=104)
13200-Anemia (Blood and lymphatic system disorders) | 65 (148)
18100-Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1)
33300-Febrile neutropenia (Blood and lymphatic system disorders) | 6 (9)
20000-Cardiac arrest (Cardiac disorders) | 1 (1)
74500-Sinus tachycardia (Cardiac disorders) | 1 (1)
28000-Ear pain (Ear and labyrinth disorders) | 1 (1)
38900-Hearing impaired (Ear and labyrinth disorders) | 9 (9)
10300-Abdominal pain (Gastrointestinal disorders) | 21 (56)
12800-Anal pain (Gastrointestinal disorders) | 1 (1)
22100-Colitis (Gastrointestinal disorders) | 1 (1)
22400-Colonic obstruction (Gastrointestinal disorders) | 1 (1)
25700-Diarrhea (Gastrointestinal disorders) | 15 (20)
27600-Dysphagia (Gastrointestinal disorders) | 1 (1)
44200-Ileal obstruction (Gastrointestinal disorders) | 1 (1)
53900-Malabsorption (Gastrointestinal disorders) | 1 (1)
55600-Mucositis oral (Gastrointestinal disorders) | 1 (1)
57600-Nausea (Gastrointestinal disorders) | 2 (2)
81900-Typhlitis (Gastrointestinal disorders) | 2 (2)
87900-Vomiting (Gastrointestinal disorders) | 4 (7)
28200-Edema face (General disorders) | 1 (1)
33900-Fever (General disorders) | 69 (204)
37200-General disorders and administration site conditions - Other (General disorders) | 1 (1)
48700-Irritability (General disorders) | 3 (3)
58600-Non-cardiac chest pain (General disorders) | 1 (2)
60600-Pain (General disorders) | 46 (134)
12000-Allergic reaction (Immune system disorders) | 9 (13)
13100-Anaphylaxis (Immune system disorders) | 9 (11)
24400-Cytokine release syndrome (Immune system disorders) | 1 (1)
20500-Catheter related infection (Infections and infestations) | 33 (63)
25600-Device related infection (Infections and infestations) | 4 (4)
29500-Enterocolitis infectious (Infections and infestations) | 3 (3)
44800-Infections and infestations - Other (Infections and infestations) | 16 (23)
53100-Lung infection (Infections and infestations) | 5 (7)
60100-Otitis media (Infections and infestations) | 2 (3)
73700-Sepsis (Infections and infestations) | 1 (1)
75200-Skin infection (Infections and infestations) | 3 (3)
76000-Small intestine infection (Infections and infestations) | 1 (1)
82300-Upper respiratory infection (Infections and infestations) | 2 (2)
83100-Urinary tract infection (Infections and infestations) | 4 (4)
86400-Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
10900-Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
11600-Alanine aminotransferase increased (Investigations) | 24 (49)
11800-Alkaline phosphatase increased (Investigations) | 2 (2)
15000-Aspartate aminotransferase increased (Investigations) | 11 (17)
17400-Blood bilirubin increased (Investigations) | 2 (6)
24100-Creatinine increased (Investigations) | 2 (2)
37500-GGT increased (Investigations) | 11 (27)
53700-Lymphocyte count decreased (Investigations) | 78 (339)
53800-Lymphocyte count increased (Investigations) | 4 (4)
58300-Neutrophil count decreased (Investigations) | 55 (193)
65800-Platelet count decreased (Investigations) | 58 (355)
83600-Urine output decreased (Investigations) | 5 (5)
88200-Weight gain (Investigations) | 2 (2)
88300-Weight loss (Investigations) | 4 (7)
88500-White blood cell decreased (Investigations) | 25 (82)
10700-Acidosis (Metabolism and nutrition disorders) | 5 (6)
13500-Anorexia (Metabolism and nutrition disorders) | 23 (25)
24700-Dehydration (Metabolism and nutrition disorders) | 5 (5)
41300-Hypercalcemia (Metabolism and nutrition disorders) | 5 (7)
41400-Hyperglycemia (Metabolism and nutrition disorders) | 11 (13)
41600-Hyperkalemia (Metabolism and nutrition disorders) | 7 (10)
41700-Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
41800-Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
42400-Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (3)
42600-Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (11)
42700-Hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
42900-Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
43100-Hypokalemia (Metabolism and nutrition disorders) | 51 (117)
43300-Hyponatremia (Metabolism and nutrition disorders) | 42 (63)
43500-Hypophosphatemia (Metabolism and nutrition disorders) | 17 (17)
16200-Back pain (Musculoskeletal and connective tissue disorders) | 10 (23)
21400-Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (3)
34200-Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
57800-Neck pain (Musculoskeletal and connective tissue disorders) | 4 (6)
60700-Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (34)
15300-Ataxia (Nervous system disorders) | 1 (1)
25300-Depressed level of consciousness (Nervous system disorders) | 1 (1)
38800-Headache (Nervous system disorders) | 6 (7)
42000-Hypersomnia (Nervous system disorders) | 1 (1)
58200-Neuralgia (Nervous system disorders) | 8 (23)
59000-Oculomotor nerve disorder (Nervous system disorders) | 1 (1)
63900-Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
64100-Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
76700-Somnolence (Nervous system disorders) | 2 (2)
11400-Agitation (Psychiatric disorders) | 4 (9)
13700-Anxiety (Psychiatric disorders) | 2 (2)
25000-Delirium (Psychiatric disorders) | 1 (1)
38500-Hallucinations (Psychiatric disorders) | 1 (1)
11100-Acute kidney injury (Renal and urinary disorders) | 1 (1)
68300-Proteinuria (Renal and urinary disorders) | 1 (2)
83000-Urinary retention (Renal and urinary disorders) | 1 (1)
14100-Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
19300-Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 (5)
23800-Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
27800-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (25)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 29 (58)
68700-Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
71600-Respiratory thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (5)
78100-Stridor (Respiratory, thoracic and mediastinal disorders) | 4 (4)
88400-Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3)
26200-Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
63600-Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
68400-Pruritus (Skin and subcutaneous tissue disorders) | 3 (6)
69700-Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
84100-Urticaria (Skin and subcutaneous tissue disorders) | 11 (22)
79000-Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1)
19800-Capillary leak syndrome (Vascular disorders) | 7 (7)
42100-Hypertension (Vascular disorders) | 4 (5)
43600-Hypotension (Vascular disorders) | 33 (67)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chimeric Antibody 14.18 With GM-CSF, IL-2 and Isotretinoin (N=104)
13200-Anemia (Blood and lymphatic system disorders) | 99 (1181)
17200-Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 (2)
18100-Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1)
25800-Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
20100-Cardiac disorders - Other (Cardiac disorders) | 6 (16)
21300-Chest pain - cardiac (Cardiac disorders) | 3 (3)
61000-Palpitations (Cardiac disorders) | 2 (2)
63100-Pericardial effusion (Cardiac disorders) | 2 (3)
74200-Sinus bradycardia (Cardiac disorders) | 7 (18)
74500-Sinus tachycardia (Cardiac disorders) | 85 (740)
78900-Supraventricular tachycardia (Cardiac disorders) | 3 (5)
81400-Tricuspid valve disease (Cardiac disorders) | 1 (1)
27900-Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 2 (2)
28000-Ear pain (Ear and labyrinth disorders) | 3 (3)
31600-External ear pain (Ear and labyrinth disorders) | 1 (1)
38900-Hearing impaired (Ear and labyrinth disorders) | 10 (10)
11200-Adrenal insufficiency (Endocrine disorders) | 1 (1)
29200-Endocrine disorders - Other (Endocrine disorders) | 1 (1)
41900-Hyperparathyroidism (Endocrine disorders) | 1 (1)
42200-Hyperthyroidism (Endocrine disorders) | 5 (5)
43400-Hypoparathyroidism (Endocrine disorders) | 1 (1)
43800-Hypothyroidism (Endocrine disorders) | 5 (7)
17800-Blurred vision (Eye disorders) | 5 (7)
23200-Conjunctivitis (Eye disorders) | 1 (1)
26000-Dry eye (Eye disorders) | 3 (3)
31900-Eye disorders - Other (Eye disorders) | 13 (14)
32100-Eye pain (Eye disorders) | 5 (5)
32200-Eyelid function disorder (Eye disorders) | 1 (1)
59300-Optic nerve disorder (Eye disorders) | 2 (2)
61900-Papilledema (Eye disorders) | 1 (1)
65600-Photophobia (Eye disorders) | 3 (3)
73200-Scleral disorder (Eye disorders) | 1 (1)
10100-Abdominal distension (Gastrointestinal disorders) | 14 (27)
10300-Abdominal pain (Gastrointestinal disorders) | 70 (284)
12800-Anal pain (Gastrointestinal disorders) | 2 (2)
17100-Bloating (Gastrointestinal disorders) | 1 (1)
21200-Cheilitis (Gastrointestinal disorders) | 10 (14)
22100-Colitis (Gastrointestinal disorders) | 1 (1)
23400-Constipation (Gastrointestinal disorders) | 36 (72)
25700-Diarrhea (Gastrointestinal disorders) | 60 (203)
26100-Dry mouth (Gastrointestinal disorders) | 3 (3)
27500-Dyspepsia (Gastrointestinal disorders) | 2 (2)
27600-Dysphagia (Gastrointestinal disorders) | 4 (4)
29400-Enterocolitis (Gastrointestinal disorders) | 4 (4)
34400-Flatulence (Gastrointestinal disorders) | 5 (7)
36400-Gastritis (Gastrointestinal disorders) | 6 (7)
36500-Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
36700-Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5 (8)
36900-Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
37600-Gingival pain (Gastrointestinal disorders) | 1 (1)
39800-Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
55600-Mucositis oral (Gastrointestinal disorders) | 3 (3)
57600-Nausea (Gastrointestinal disorders) | 55 (188)
59700-Oral pain (Gastrointestinal disorders) | 4 (4)
70800-Rectal ulcer (Gastrointestinal disorders) | 1 (1)
77900-Stomach pain (Gastrointestinal disorders) | 7 (13)
80200-Toothache (Gastrointestinal disorders) | 2 (2)
87900-Vomiting (Gastrointestinal disorders) | 65 (309)
21500-Chills (General disorders) | 21 (34)
28200-Edema face (General disorders) | 56 (110)
28300-Edema limbs (General disorders) | 36 (61)
28400-Edema trunk (General disorders) | 5 (6)
32500-Facial pain (General disorders) | 2 (2)
33200-Fatigue (General disorders) | 34 (73)
33900-Fever (General disorders) | 102 (1117)
34600-Flu like symptoms (General disorders) | 2 (7)
35000-Gait disturbance (General disorders) | 3 (5)
37200-General disorders and administration site conditions - Other (General disorders) | 4 (7)
43700-Hypothermia (General disorders) | 1 (2)
45000-Infusion related reaction (General disorders) | 4 (10)
45200-Injection site reaction (General disorders) | 16 (23)
48700-Irritability (General disorders) | 33 (74)
52800-Localized edema (General disorders) | 10 (14)
54000-Malaise (General disorders) | 4 (4)
58600-Non-cardiac chest pain (General disorders) | 6 (7)
60600-Pain (General disorders) | 82 (746)
12000-Allergic reaction (Immune system disorders) | 33 (123)
24400-Cytokine release syndrome (Immune system disorders) | 2 (2)
18800-Bronchial infection (Infections and infestations) | 1 (1)
20500-Catheter related infection (Infections and infestations) | 5 (6)
23300-Conjunctivitis infective (Infections and infestations) | 1 (1)
29500-Enterocolitis infectious (Infections and infestations) | 9 (13)
30400-Esophageal infection (Infections and infestations) | 1 (1)
44800-Infections and infestations - Other (Infections and infestations) | 21 (28)
53100-Lung infection (Infections and infestations) | 3 (3)
55500-Mucosal infection (Infections and infestations) | 1 (1)
57200-Nail infection (Infections and infestations) | 1 (1)
60100-Otitis media (Infections and infestations) | 4 (5)
62000-Papulopustular rash (Infections and infestations) | 1 (1)
62200-Paronychia (Infections and infestations) | 1 (3)
65200-Pharyngitis (Infections and infestations) | 3 (5)
72600-Rhinitis infective (Infections and infestations) | 3 (4)
74600-Sinusitis (Infections and infestations) | 2 (2)
75200-Skin infection (Infections and infestations) | 6 (8)
76000-Small intestine infection (Infections and infestations) | 1 (1)
82300-Upper respiratory infection (Infections and infestations) | 9 (11)
83100-Urinary tract infection (Infections and infestations) | 6 (8)
19400-Bruising (Injury, poisoning and procedural complications) | 8 (9)
25500-Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2)
45700-Injury poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 2 (3)
66800-Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
86400-Vascular access complication (Injury, poisoning and procedural complications) | 8 (13)
10900-Activated partial thromboplastin time prolonged (Investigations) | 8 (10)
11600-Alanine aminotransferase increased (Investigations) | 90 (507)
11800-Alkaline phosphatase increased (Investigations) | 20 (64)
15000-Aspartate aminotransferase increased (Investigations) | 91 (399)
17400-Blood bilirubin increased (Investigations) | 15 (40)
21700-Cholesterol high (Investigations) | 3 (3)
24100-Creatinine increased (Investigations) | 31 (137)
28700-Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
37500-GGT increased (Investigations) | 20 (87)
39400-Hemoglobin increased (Investigations) | 9 (29)
45800-INR increased (Investigations) | 5 (5)
48400-Investigations - Other (Investigations) | 3 (6)
53700-Lymphocyte count decreased (Investigations) | 87 (904)
53800-Lymphocyte count increased (Investigations) | 4 (4)
58300-Neutrophil count decreased (Investigations) | 67 (376)
65800-Platelet count decreased (Investigations) | 97 (780)
88200-Weight gain (Investigations) | 56 (227)
88300-Weight loss (Investigations) | 21 (54)
88500-White blood cell decreased (Investigations) | 89 (737)
10700-Acidosis (Metabolism and nutrition disorders) | 3 (10)
13500-Anorexia (Metabolism and nutrition disorders) | 32 (84)
24700-Dehydration (Metabolism and nutrition disorders) | 13 (16)
41300-Hypercalcemia (Metabolism and nutrition disorders) | 26 (48)
41400-Hyperglycemia (Metabolism and nutrition disorders) | 61 (195)
41600-Hyperkalemia (Metabolism and nutrition disorders) | 35 (71)
41700-Hypermagnesemia (Metabolism and nutrition disorders) | 17 (52)
41800-Hypernatremia (Metabolism and nutrition disorders) | 12 (18)
42400-Hypertriglyceridemia (Metabolism and nutrition disorders) | 84 (205)
42500-Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
42600-Hypoalbuminemia (Metabolism and nutrition disorders) | 101 (890)
42700-Hypocalcemia (Metabolism and nutrition disorders) | 96 (579)
42900-Hypoglycemia (Metabolism and nutrition disorders) | 43 (95)
43100-Hypokalemia (Metabolism and nutrition disorders) | 85 (392)
43200-Hypomagnesemia (Metabolism and nutrition disorders) | 41 (119)
43300-Hyponatremia (Metabolism and nutrition disorders) | 95 (524)
43500-Hypophosphatemia (Metabolism and nutrition disorders) | 69 (211)
54900-Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2 (5)
14700-Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
16200-Back pain (Musculoskeletal and connective tissue disorders) | 25 (70)
18200-Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
19700-Buttock pain (Musculoskeletal and connective tissue disorders) | 4 (4)
21400-Chest wall pain (Musculoskeletal and connective tissue disorders) | 6 (22)
37300-Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
49800-Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
55900-Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
56300-Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 (6)
56500-Myalgia (Musculoskeletal and connective tissue disorders) | 10 (11)
57800-Neck pain (Musculoskeletal and connective tissue disorders) | 14 (32)
60700-Pain in extremity (Musculoskeletal and connective tissue disorders) | 48 (155)
11500-Akathisia (Nervous system disorders) | 2 (2)
22000-Cognitive disturbance (Nervous system disorders) | 1 (1)
22800-Concentration impairment (Nervous system disorders) | 1 (1)
25300-Depressed level of consciousness (Nervous system disorders) | 1 (1)
25900-Dizziness (Nervous system disorders) | 3 (5)
38800-Headache (Nervous system disorders) | 31 (76)
42000-Hypersomnia (Nervous system disorders) | 1 (1)
51800-Lethargy (Nervous system disorders) | 5 (5)
54400-Memory impairment (Nervous system disorders) | 1 (1)
54500-Meningismus (Nervous system disorders) | 1 (2)
55400-Movements involuntary (Nervous system disorders) | 4 (4)
58100-Nervous system disorders - Other (Nervous system disorders) | 2 (3)
58200-Neuralgia (Nervous system disorders) | 5 (13)
58700-Nystagmus (Nervous system disorders) | 1 (1)
59000-Oculomotor nerve disorder (Nervous system disorders) | 1 (1)
62100-Paresthesia (Nervous system disorders) | 2 (2)
64100-Peripheral sensory neuropathy (Nervous system disorders) | 11 (16)
73600-Seizure (Nervous system disorders) | 2 (2)
76700-Somnolence (Nervous system disorders) | 7 (7)
81300-Tremor (Nervous system disorders) | 3 (3)
67200-Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1)
11400-Agitation (Psychiatric disorders) | 24 (40)
13700-Anxiety (Psychiatric disorders) | 14 (23)
23000-Confusion (Psychiatric disorders) | 7 (10)
25400-Depression (Psychiatric disorders) | 3 (6)
38500-Hallucinations (Psychiatric disorders) | 10 (14)
45900-Insomnia (Psychiatric disorders) | 7 (8)
54100-Mania (Psychiatric disorders) | 1 (1)
68500-Psychiatric disorders - Other (Psychiatric disorders) | 3 (3)
71700-Restlessness (Psychiatric disorders) | 4 (6)
11100-Acute kidney injury (Renal and urinary disorders) | 2 (3)
21800-Chronic kidney disease (Renal and urinary disorders) | 1 (1)
39300-Hematuria (Renal and urinary disorders) | 36 (93)
68300-Proteinuria (Renal and urinary disorders) | 43 (144)
71000-Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (4)
82800-Urinary frequency (Renal and urinary disorders) | 1 (1)
82900-Urinary incontinence (Renal and urinary disorders) | 1 (1)
83000-Urinary retention (Renal and urinary disorders) | 30 (63)
83300-Urinary tract pain (Renal and urinary disorders) | 4 (9)
83400-Urinary urgency (Renal and urinary disorders) | 1 (1)
83500-Urine discoloration (Renal and urinary disorders) | 5 (13)
37400-Genital edema (Reproductive system and breast disorders) | 1 (4)
62600-Pelvic pain (Reproductive system and breast disorders) | 1 (1)
62900-Penile pain (Reproductive system and breast disorders) | 2 (3)
71400-Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 (3)
85600-Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
12100-Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 15 (18)
15400-Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 (9)
19000-Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 2 (2)
19300-Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 10 (16)
23800-Cough (Respiratory, thoracic and mediastinal disorders) | 74 (220)
27800-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (11)
29700-Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6)
40700-Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
41000-Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 32 (99)
51500-Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
51600-Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
57500-Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 23 (39)
65300-Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
65900-Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
66200-Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (3)
66300-Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
66700-Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
67600-Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
68700-Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
71600-Respiratory thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 34 (242)
72200-Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
76200-Sneezing (Respiratory, thoracic and mediastinal disorders) | 6 (6)
76800-Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 (12)
88400-Wheezing (Respiratory, thoracic and mediastinal disorders) | 17 (37)
12200-Alopecia (Skin and subcutaneous tissue disorders) | 28 (36)
19500-Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
26200-Dry skin (Skin and subcutaneous tissue disorders) | 69 (175)
29900-Erythema multiforme (Skin and subcutaneous tissue disorders) | 8 (11)
42300-Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
57300-Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
60900-Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
63600-Periorbital edema (Skin and subcutaneous tissue disorders) | 16 (27)
65700-Photosensitivity (Skin and subcutaneous tissue disorders) | 2 (2)
68400-Pruritus (Skin and subcutaneous tissue disorders) | 62 (223)
69600-Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (6)
69700-Rash maculo-papular (Skin and subcutaneous tissue disorders) | 58 (130)
74700-Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 20 (51)
74800-Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
74900-Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
75000-Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (4)
75100-Skin induration (Skin and subcutaneous tissue disorders) | 3 (3)
75300-Skin ulceration (Skin and subcutaneous tissue disorders) | 4 (4)
84100-Urticaria (Skin and subcutaneous tissue disorders) | 46 (139)
19800-Capillary leak syndrome (Vascular disorders) | 53 (131)
34700-Flushing (Vascular disorders) | 8 (10)
41100-Hot flashes (Vascular disorders) | 2 (2)
42100-Hypertension (Vascular disorders) | 56 (406)
43600-Hypotension (Vascular disorders) | 81 (768)
79600-Thromboembolic event (Vascular disorders) | 1 (1)
86500-Vascular disorders - Other (Vascular disorders) | 3 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less